CLINICAL TRIAL: NCT06039397
Title: The Effect of Semi Fowler 30' Right Lateral on Cardiac Output in Acute Heart Failure
Acronym: SETTLECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Ryan Budiyanto, Clinical Investigator, Indonesia University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 01.202303.046
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Output, High; Heart Failure; Pulmonary Edema With Heart Failure; Dyspnea; Cardiac; Arrythmia
Keywords: Cardiac Output; Heart Failure; Body Positioning; Right Lateral Body Position; Semifowler
MeSH Terms: conditions — Cardiac Output, High; Heart Failure; Dyspnea; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-fowler 30" Right Lateral (Experimental)
  Interventions: Behavioral: Semifowler 30' Right Lateral Body Position
- Conventional care (Active Comparator)
  Interventions: Behavioral: Semifowler 30' Right Lateral Body Position

INTERVENTIONS:
Behavioral: Semifowler 30' Right Lateral Body Position — Semifowler 30' Right Lateral Body Position Is a regulation of body position by placing the patient's body in a semi-fowler and lateral resting position of 30 degrees

SUMMARY:
Heart failure is a special clinical syndrome such as difficulty breathing, fatigue, and swollen legs characterized by increased JVP, crackle lung sounds, and peripheral edema caused by heart disorders both structural and/or functional, resulting in decreased cardiac output and increased intracardiac pressure at rest and activity. Body positioning has been shown to affect stroke volume and parasympathetic modulating activity. The right lateral 30" semifowler position is a very safe position in heart failure patients admitted to the ICU. Although body positioning can affect stroke volume, and parasympathetic modulation, it is not yet clear what effect it has on cardiac output

ELIGIBILITY:
Inclusion Criteria:

* The patient was diagnosed with acute decompensated heart failure,
* fully conscious,
* not intubated,
* >18 years old,
* had no mobility problems,
* palpable radial artery pulsation,
* was not under the influence of anti-hypotensive drugs,
* willing to be a respondent,
* LVEF <50%.

Exclusion Criteria:

* Pulmonary edema,
* severe valve disease comorbidities,
* receiving high doses of anti-hypotensive treatment,
* heart failure readmission in the last 3 months,
* finger edema,
* use of mechanical circulatory support,
* irregular rhythms,
* artificial pacemaker attached,
* obesity
* peripheral perfusion disorders
* cardiogenic shock

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | 15 Minutes
  The amount of blood volume pumped by the heart for 1 minute in liters

CONTACTS AND LOCATIONS:
Locations (1):
- Ryan Budiyanto, Jakarta, West Jakarta, Indonesia

REFERENCES:
- [Background] Gottlieb LA, Blanco LSY, Hocini M, Dekker LRC, Coronel R. Self-Reported Onset of Paroxysmal Atrial Fibrillation Is Related to Sleeping Body Position. Front Physiol. 2021 Jul 15;12:708650. doi: 10.3389/fphys.2021.708650. eCollection 2021. PMID 34335312
- [Background] Carlisle MA, Fudim M, DeVore AD, Piccini JP. Heart Failure and Atrial Fibrillation, Like Fire and Fury. JACC Heart Fail. 2019 Jun;7(6):447-456. doi: 10.1016/j.jchf.2019.03.005. PMID 31146871
- [Background] Chen GY, Kuo CD. The effect of the lateral decubitus position on vagal tone. Anaesthesia. 1997 Jul;52(7):653-7. doi: 10.1111/j.1365-2044.1997.114-az0106.x. PMID 9244024
- [Result] Miyamoto S, Fujita M, Sekiguchi H, Okano Y, Nagaya N, Ueda K, Tamaki S, Nohara R, Eiho S, Sasayama S. Effects of posture on cardiac autonomic nervous activity in patients with congestive heart failure. J Am Coll Cardiol. 2001 Jun 1;37(7):1788-93. doi: 10.1016/s0735-1097(01)01249-9. PMID 11401112
- [Result] Pan H, Xu Z, Yan H, Gao Y, Chen Z, Song J, Zhang Y. Lying position classification based on ECG waveform and random forest during sleep in healthy people. Biomed Eng Online. 2018 Aug 30;17(1):116. doi: 10.1186/s12938-018-0548-7. PMID 30165874
- See also: Effect of right lateral position on hemodynamics and comfort of patients with heart failure at Harapan Kita — https://www.lontar.ui.ac.id/detail?id=20390020&lokasi=lokal